CLINICAL TRIAL: NCT07350486
Title: A Cluster-Randomized Trial of Large Language Model-Enabled Coordinated Management for Hypertension, Diabetes, and Dyslipidemia in Community Settings (LLM-CoManage Trial)
Brief Title: LLM-CoManage: Large Language Model-Enabled Co-Management of Hypertension, Diabetes, and Dyslipidemia
Acronym: LLM-CoManage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Hospital of China Medical University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Zhejiang University (Other); Shandong Provincial Hospital (Other Government); Cangzhou Central Hospital (Other)
Responsible Party: Principal Investigator, Yingxian Sun, Chief of Department of Cardiology in First Hospital of China Medical University, First Hospital of China Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMU-HyperMindRCT-2025
Record Dates: First submitted 2025-12-25; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Diabetes; Dyslipidemia
Keywords: Large Language Model; Co-Management
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome Assessment Committee members will be blinded to outcome assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLM-Enabled Intervention Group (Active Comparator): LLM-enabled community physicians delivered integrated, guideline-based management
  Interventions: Other: LLM-Enabled Clinician-Patient Co-management
- Usual Care Control Group (No Intervention): Community physicians provided routine care according to local primary health service standards

INTERVENTIONS:
Other: LLM-Enabled Clinician-Patient Co-management — The intervention is a LLM-enabled, community-based integrated management strategy for cardiometabolic multimorbidity. The LLM system functions as the central intelligence layer, integrating multi-condition clinical information, delivering real-time decision support, coordinating care workflows, and facilitating continuous patient engagement. Within this LLM-enabled framework, community physicians-after standardized training-serve as the core executors of care, delivering guideline-based pharmacologic treatment, lifestyle counseling, and structured monitoring of coexisting cardiometabolic conditions. Policy-aligned performance incentives are used to support physician engagement and implementation fidelity, without altering medication access or underlying clinical protocols.
  The LLM-enabled intervention is implemented through the HyperMind system, an integrated platform that simultaneously supports clinicians, patients, and health-system oversight.
  Arms: LLM-Enabled Intervention Group

SUMMARY:
This study aims to evaluate the effectiveness of a large language model (LLM)-supported, community-based integrated management model in improving cardiometabolic multimorbidity control among adults with hypertension and coexisting diabetes or dyslipidemia. Adopting an interventional study design, eligible patients will be recruited to compare the disease control indicators between LLM-assisted management and conventional management, so as to verify the effectiveness and safety of the former.

ELIGIBILITY:
Inclusion Criteria:

Participating communities must meet all of the following criteria:

* Have a designated community physician responsible for primary care who is capable of using a smartphone with stable internet access for clinical communication and LLM-assisted management;
* No plan for administrative merger or restructuring within the next three years;
* Located at least 2 kilometers away from adjacent participating communities (to minimize contamination between clusters).

Eligible participants must fulfill all of the following conditions:

* Aged 40 years or older;
* Uncontrolled hypertension, defined as systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg;
* Coexisting diabetes (HbA1c ≥ 7.0%) or coexisting dyslipidemia (LDL-C ≥ 3.4 mmol/L[130 mg/dL]);
* Able to use a smartphone independently or with assistance from family members;
* Has resided in the participating community for at least 6 months;
* Has no plan to relocate in the next 3 years;
* Enrolled in basic medical insurance for urban and rural residents, employee medical insurance, or the New Rural Cooperative Medical Scheme;
* Not currently pregnant or planning pregnancy during the study period;
* Free from malignant tumors and deemed to have a life expectancy of at least 3 years, as judged by study physicians;
* Willing and able to provide written informed consent.

Exclusion Criteria:No specific exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The between-group difference in the proportion of participants achieving simultaneous control of hypertension and either diabetes or dyslipidemia. | 6 months after baseline
  Simultaneous control is defined as BP < 130/80 mmHg and at least one of the following: HbA1c < 7.0% or LDL-C < 2.6 mmol/L (100 mg/dL), with a stricter threshold of < 1.9 mmol/L (70 mg/dL) for participants with cardiovascular disease(CVD).

SECONDARY OUTCOMES:
Proportion of participants achieving control of individual risk factors: BP < 130/80 mmHg (or < 140/90 mmHg); HbA1c < 7.0%; and LDL-C < 2.6 mmol/L (100 mg/dL) or < 1.9 mmol/L (70 mg/dL) for those with CVD. | 6 months after baseline
  The proportion of participants achieving target control of each individual risk factor, including blood pressure, HbA1c, and LDL-C.
Mean systolic blood pressure changes. | 6 months after baseline
  Mean systolic blood pressure changes of participants.
Mean diastolic blood pressure changes. | 6 months after baseline.
  Mean diastolic blood pressure changes of participants.
Mean HbA1c changes. | 6 months after baseline.
  Mean HbA1c changes of participants.
Mean LDL-C changes. | 6 months after baseline.
  Mean LDL-C changes of participants.
Proportion of participants achieving simultaneous control of BP, HbA1c, and LDL-C. | 6 months after baseline
  The proportion of participants achieving simultaneous control of blood pressure, HbA1c, and LDL-C.
Awareness and treatment rates for hypertension, diabetes, and dyslipidemia. | 6 months after baseline
  Rates of disease awareness and treatment for hypertension, diabetes, and dyslipidemia.
Proportion of participants receiving integrated, guideline-based management of all indicated conditions. | 6 months after baseline
  The proportion of participants receiving integrated, guideline-based management for indicated conditions.
Mean health expenditures and within-trial cost-utility. | 6 months after baseline
  Mean health care expenditures and within-trial cost-utility outcomes.
Net changes in estimated 10-year risk for atherosclerotic CVD. | 6 months after baseline
  Net change in estimated 10-year atherosclerotic cardiovascular disease risk.
Changes in treatment adherence. | 6 months after baseline
  Change in treatment adherence among participants.
Improvements in behavioral risk factors (e.g., diet, physical activity, tobacco use, lifestyle intervention uptake). | 6 months after baseline
  Changes in behavioral risk factors including diet, physical activity, and tobacco use.
Patient-reported outcomes related to satisfaction. | 6 months after baseline
  Patient-reported satisfaction with LLM will be assessed using a structured scale.
Patient-reported outcomes related to self-management. | 6 months after baseline.
  Patient-reported self-management will be assessed using a structured scale.
Patient-reported outcomes related to quality of life. | 6 months after baseline.
  Patient-reported quality of life will be assessed using a structured scale.
Adoption and utilization of the LLM system by physicians and patients. | 6 months after baseline
  The extent of physician and patient adoption and use of the LLM-based system.
Patterns of AI-assisted recommendations and digital interactions. | 6 months after baseline
  The patterns of Artificial Intelligence(AI)-assisted recommendations and related digital interactions generated during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, MD, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided